CLINICAL TRIAL: NCT06730178
Title: Calo Psychiatric Center
Brief Title: Using Generalized Estimating Equation Analysis in a Study of Relaxation Training in Patients With Insomnia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Calo Psychiatric Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9802
Record Dates: First submitted 2024-12-08; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Sleep Disorder; Insomnia Type
Keywords: Insomnia; Relaxation Training; Generalized Estimating Equation
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Initiation and Maintenance Disorders | interventions — Relaxation Therapy

STUDY DESIGN:
Intervention Model Description: All insomnia patients were asked to complete the insomnia scales. The goals and processes of relaxation training were explained by therapists. The patients were asked to record data before relaxation training, inclusive of all sleep durations, the frequency of night waking, the time needed to fall asleep, and medication history. The insomnia scales were completed again one week later, and the relaxation training started in the second week. The patients recorded their sleep conditions every day and underwent relaxation training intervention for 4 weeks. They were treated similarly, four times in total.
Masking Description: Of 47 qualified subjects, 24 volunteers took part in this study after the researchers had explained the study process. All subjects had been diagnosed as having primary insomnia or insomnia related to medical and psychiatric comorbid diagnoses using the D Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) diagnostic criteria.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Relaxation training in patients with insomnia (Experimental): The goals and processes of relaxation training were explained by therapists. The patients were asked to record data before relaxation training, inclusive of all sleep durations, the frequency of night waking, the time needed to fall asleep, and medication history. The insomnia scales were completed again one week later, and the relaxation training started in the second week. The patients recorded their sleep conditions every day and underwent relaxation training intervention for 4 weeks.
  Interventions: Behavioral: relaxation training

INTERVENTIONS:
Behavioral: relaxation training — The training tapes used were meditation relaxation training tapes translated form Jacobson progressive relaxation technique with copyrights. The tapes were recorded by a male therapist. Participants were instructed to perform the treatment in the evening, preferably just before bedtime, total time was 15 minutes.

SUMMARY:
Background: The purpose of this study was to examine the improvement in insomnia patients using Relaxation Training, and to use the Generalized Estimating Equation model (GEE-I) to analyze the results of repeated measurements and observe the difference between the subjective perception and the objective measurement of sleep duration.

Methods: There were 24 subjects diagnosed as insomnia who completed the treatment course and 5 times evaluation. Of the 24 subjects, 7 accepted the sleep electroencephalogram (EEG). Relaxation training shortened the duration of sleep onset time and decreased the frequency of night awakening.

DETAILED DESCRIPTION:
Of 47 qualified subjects, 24 volunteers took part in this study after the researchers had explained the study process.The patients were asked to keep a sleep diary. In the diaries, they recorded the time they went to bed and fell asleep, the duration to sleep onset (from "go to the bed" to "fall asleep"), the frequency of night waking, the time of getting up, and any medication history. Patients were instructed to perform the treatment in the evening, preferably just before bedtime, total time was 15 minutes.The patients recorded their sleep conditions every day and underwent relaxation training intervention for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* All subjects had been diagnosed as having primary insomnia or insomnia related to medical and psychiatric comorbid diagnoses using the D Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) diagnostic criteria.

Exclusion Criteria:

* Patients who had comorbid serious medical illnesses, and pregnant and lactating women were excluded.

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2009-10-30 (Actual); Study Completion 2009-10-30 (Actual)

PRIMARY OUTCOMES:
the improvement of relaxation training tape | 4 weeks
  Participants were instructed to perform the treatment in the evening, preferably just before bedtime, total time was 15 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: For-Wey Lung, MD, ScD, Principal Investigator — Calo Psychiatric Center

IPD SHARING:
Plan to Share IPD: No
The data in this study are available to other researchers upon request.